CLINICAL TRIAL: NCT04597138
Title: The Relationship Between Deep Venous Thrombus Characteristics and Venous Dynamics With Subsequent Thrombus Resolution and Post-thrombotic Syndrome
Brief Title: Deep Venous Thrombus Characteristics and Venous Dynamics With Subsequent Thrombus Resolution and Post-thrombotic Syndrome
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Damon E. Houghton, Principal Investigator, Mayo Clinic
Other Study IDs: 20-002573
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Deep Vein Thrombosis
Keywords: Thrombus Resolution; Post-Thrombotic Syndrome
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to examine in vivo thrombosis characteristics with ultrasound shear wave elastography (SWE) and determine the relationship with thrombus resolution and postthrombotic syndrome (PTS) in patients with acute proximal Deep Vein Thrombosis (DVT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute, proximal (popliteal and above) DVT with or without Pulmonary Embolism within 72 hours
* ≥18 Years Old

Exclusion Criteria

* prior episode of DVT
* contraindication to standard therapeutic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute, proximal DVT initiating anticoagulation
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Thrombus Resolution | 3 Months after diagnosis of DVT.
  Ultrasound images of lower extremity DVTs comparing the initial diagnostic image of thrombus to a subsequent study performed after 3 months of anticoagulation.The lower extremity venous system is divided into 12 segments. Each vein segment will be analyzed on initial ultrasound and recorded 0 (no DVT), 1 (non-occlusive DVT), or 2 (occlusive DVT). The follow up ultrasound will be analyzed per vein segment and recorded as no residual thrombus, minimal chronic post-thrombotic changes, > 50% resolution, < 50% resolution, near occlusive DVT, no change, and progressive DVT.

SECONDARY OUTCOMES:
Post-thrombotic syndrome | 6 months after diagnosis of DVT
  Measured using the Villalta Score. Scale 0-33 with higher values indicating more severe symptoms.
Vein Specific Quality of Life | 6 months after diagnosis of DVT
  Measured using The Venous Insufficiency Epidemiological and Economic Study (VEINES) QOL survey. Scores range from 0-100 with higher scores indicating better quality of life.

OTHER OUTCOMES:
Post-thrombotic syndrome | 3 and 12 months after diagnosis of DVT
  Measured using the Villalta Score. Scale 0-33 with higher values indicating more severe symptoms.
Vein Specific Quality of Life | 3 and 12 months after diagnosis of DVT
  Measured using The Venous Insufficiency Epidemiological and Economic Study (VEINES) QOL survey. Scores range from 0-100 with higher scores indicating better quality of life.
Thrombus Resolution | 3 Months after diagnosis of DVT.
  Measured quantitatively by outflow parameters on air plethysmography with expelled volume measured at 1 second x 60 sec (ml/100ml/minute), expelled volume after 4 seconds, and maximum volume expelled.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Houghton, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials